CLINICAL TRIAL: NCT01823510
Title: Comparative Study of the Antithrombotic Effects of Ticagrelor and Clopidogrel in Type 2 Diabetic Patients
Brief Title: Ticagrelor Versus Clopidogrel in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Juan J Badimon (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Juan J Badimon, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 13-0208
Record Dates: First submitted 2013-03-29; First posted 2013-04-04 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Type-2 Diabetes Mellitus; Coronary Artery Disease
Keywords: Antiplatelet; Ticagrelor; Clopidogrel; Thrombosis; Diabetes; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease; Thrombosis; Diabetes Mellitus | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor + Aspirin (Experimental): Loading-dose plus daily-dosing for 5-7 days.
  Interventions: Drug: Ticagrelor + Aspirin
- Clopidogrel + Aspirin (Active Comparator): Loading-dose plus daily-dosing for 5-7 days.
  Interventions: Drug: Clopidogrel + Aspirin

INTERVENTIONS:
Drug: Ticagrelor + Aspirin — Single loading doses of Ticagrelor (180 mg) and ASA (325 mg), followed by daily dosing for 5-7 days (ticagrelor 90 mg twice daily + ASA 81 mg once daily).
  Other Names: Brilinta (ticagrelor); Aspirin (ASA)
  Arms: Ticagrelor + Aspirin
Drug: Clopidogrel + Aspirin — Single loading doses of Clopidogrel (600 mg) and ASA (325 mg), followed by daily dosing for 5-7 days (clopidogrel 75 mg + ASA 81 mg once daily).
  Other Names: Plavix (clopidogrel); Aspirin (ASA)
  Arms: Clopidogrel + Aspirin

SUMMARY:
The purpose of this study is to determine whether treatment with ticagrelor + aspirin is more effective than treatment with clopidogrel + aspirin in patients with type-2 diabetes. Both treatments will be given (separately) to all subjects as a one-time loading dose (i.e. higher than a normal daily dose), followed by daily dose for the next 5 to 7 days. Effectiveness of treatment will be measured with specialized blood tests before the loading dose, at two time-points after the loading dose, and once after the last daily dose.

DETAILED DESCRIPTION:
The rising prevalence of diabetes mellitus and its associated cardiovascular complications present a major burden to healthcare providers worldwide. Cardiovascular mortality is much higher among subjects with Type 2 Diabetes Mellitus (T2DM). Increased platelet reactivity is considered a potential link between the two diseases. Thus, given the higher blood thrombogenicity of T2DM with CAD, the availability of more potent antiplatelet drugs should be associated with improvements in the prevention of cardiovascular events in the diabetic populations. Ticagrelor has been shown to possess a faster onset of action and more potency than clopidogrel. Furthermore, the PLATO has shown that these characteristics results in a significant reduction in Cardiovascular events and even death as compared with Clopidogrel.

We plan to compare the antithrombotic activity of ticagrelor versus clopidogrel in T2DM patients using a cross-over study design. Each participant will be randomly assigned to receive ticagrelor/clopidogrel + aspirin as a loading dose followed by 5-7 days of daily maintenance dosing. After a washout period of 1-2 weeks, each participant will receive the second treatment (clopidogrel/ticagrelor + aspirin) again as a loading dose followed by 5-7 days of daily dosing. Platelet function will be tested at pre-treatment baseline, two post-dose time-points on the day of loading dose, and one time-point after the last maintenance dose on day 5-7. Platelet testing will be carried out using the following methodologies:

1. Badimon Perfusion Chamber: an ex-vivo model of thrombosis that has been extensively utilized for evaluation of antithrombotic or prothrombotic effects under various pathological states. The model involves native blood perfusing over a thrombogenic substrate, triggering thrombus formation that can be measured by planimetry.
2. Platelet Aggregation - Multiplate Analyzer.
3. Platelet Aggregation - VerifyNow P2Y12 assay.
4. Vasodilator-Stimulated Phosphoprotein (VASP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type-2 diabetes being treated with oral or parenteral hypoglycemic therapy or both.
* Have not had thienopyridine therapy for at least 30 days before the study.
* Are of legal age (at least 18 years of age but less than 75 years of age) and competent mental condition to provide written informed consent.
* For women of child-bearing potential only test negative for pregnancy at the time of enrollment.

Exclusion Criteria:

* Have a defined need for thienopyridine therapy.
* Subjects within ≤30 days of coronary artery bypass graft (CABG) surgery or percutaneous coronary intervention (PCI).
* Known glycosylated hemoglobin (HbA1c) ≥10 mg/dL within last 3 months prior to study entry.
* Have received fibrinolytic therapy <48 hours prior to randomization.
* Have active internal bleeding or history of bleeding diathesis.
* Have clinical findings that are, in the judgment of the investigator, associated with an increased risk of bleeding.
* Have history of ischemic or hemorrhagic stroke, transient ischemic attack (TIA) or intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Have an International Normalized Ratio (INR) known to be >1.5 within 1 week of study entry.
* Have a known platelet count of <100,000/mm3 within 1 week of study entry.
* Have known anemia (hemoglobin [Hgb] <10 gm/dL) within 1 week of study entry.
* Are receiving or will receive oral anticoagulation or other antiplatelet therapy (other than ASA) that cannot be safely discontinued for the duration of the trial.
* Are receiving daily treatment with non-steroidal anti-inflammatory drugs (NSAIDS) that cannot be discontinued.
* Have a concomitant medical illness that in the opinion of the investigator may interfere with or prevent completion in this study.
* Have known severe hepatic dysfunction (e.g., cirrhosis or portal hypertension).
* Have a history of intolerance or allergy to ASA or approved thienopyridines (ticlopidine or clopidogrel).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Badimon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Zafar MU, Baber U, Smith DA, Sartori S, Contreras J, Rey-Mendoza J, Linares-Koloffon CA, Escolar G, Mehran R, Fuster V, Badimon JJ. Antithrombotic potency of ticagrelor versus clopidogrel in type-2 diabetic patients with cardiovascular disease. Thromb Haemost. 2017 Oct 5;117(10):1981-1988. doi: 10.1160/TH17-04-0277. Epub 2017 Aug 24. PMID 28837213

RESULTS

PARTICIPANT FLOW:
Groups:
- Tica-Clop: Participants received Ticagrelor plus ASA (loading-dose plus daily-dose for 5-7 days), followed by Washout (14 days), and then Clopidogrel plus ASA (loading-dose plus daily-dose for 5-7 days).
- Clop-Tica: Participants received Clopidogrel plus ASA (loading-dose plus daily-dose for 5-7 days), followed by Washout (14 days), and then Ticagrelor plus ASA (loading-dose plus daily-dose for 5-7 days).
Period: Days 1-7
Arm/Group | Tica-Clop | Clop-Tica
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Days 8-21
Arm/Group | Tica-Clop | Clop-Tica
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Days 22-28
Arm/Group | Tica-Clop | Clop-Tica
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Type 2 Diabetic Patients: All participants receive both Ticagrelor and Clopidogrel (each with aspirin) in a cross-over design. Treatment sequence (Tica-Clop OR Clop-Tica) was randomly assigned and with a 2-week washout period in between (i.e., "Tica/Clop (5-7 days)", "Washout (14 days)", and "Clop/Tica (5-7 days)").
Arm/Group | Type 2 Diabetic Patients
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.9 (4.5)
Diabetes, type-2 [Count of Participants; unit: Participants] | 20
Hypertension [Count of Participants; unit: Participants] | 17
Hypercholesterolemia [Count of Participants; unit: Participants] | 19
Smoking [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Thrombus Formation
Description: Thrombus formation in Badimon Perfusion Chamber high-shear) (ex vivo model of thrombosis).
Time Frame: up to 7 days
Measure: Mean (Standard Error); unit: percentage of baseline size
Arm/Group | Ticagrelor + Aspirin | Clopidogrel + Aspirin
Number analyzed (Participants) | 20 | 20
percentage of baseline size
  2 hour post loading dose | 66.9 (8.0) | 84.4 (6.4)
  6 hours post loading dose | 59.9 (8.0) | 79.8 (6.4)
  5-7 days of maintenance dose | 68.9 (8.3) | 82.6 (6.5)

2. Secondary Outcome: Platelet Reactivity
Description: Platelet reactivity by Multiplate Analyzer
Time Frame: up to 7 days
Measure: Mean (Standard Error); unit: percentage of baseline Unit
Arm/Group | Ticagrelor + Aspirin | Clopidogrel + Aspirin
Number analyzed (Participants) | 20 | 20
percentage of baseline Unit
  2 hour post-loading dose | 20.5 (7.4) | 54.5 (14.4)
  6 hour post-loading dose | 20.6 (7.5) | 43.6 (14.6)
  5-7 days of maintenance dosing | 24.2 (7.7) | 45.5 (14.4)

3. Secondary Outcome: P2Y12 Reaction Unit (PRU)
Description: Platelet reactivity by measuring P2Y12 Reaction Unit using Accumetrics VerifyNow
Time Frame: up to 7 days
Measure: Mean (Standard Error); unit: percentage of baseline PRU
Arm/Group | Ticagrelor + Aspirin | Clopidogrel + Aspirin
Number analyzed (Participants) | 20 | 20
percentage of baseline PRU
  2 hour post-loading dose | 14.8 (7.2) | 77.8 (11.8)
  6 hour post-loading dose | 8.2 (7.5) | 66.8 (11.9)
  5-7 days of maintenance dosing | 14.5 (7.5) | 62.7 (11.8)

4. Secondary Outcome: Platelet Reactivity Index (PRI)
Description: Platelet reactivity index by Vasodilator-Stimulated Phosphoprotein phosphorylation (VASP) assay.
Time Frame: up to 7 days
Measure: Mean (Standard Error); unit: percentage of baseline PRI
Arm/Group | Ticagrelor + Aspirin | Clopidogrel + Aspirin
Number analyzed (Participants) | 20 | 20
percentage of baseline PRI
  2 hour post-loading dose | 21.8 (2.5) | 85.8 (3.3)
  6 hour post-loading dose | 17.8 (2.5) | 82.5 (3.4)
  5-7 days of maintenance dosing | 17.2 (2.5) | 68.4 (3.4)

ADVERSE EVENTS:
Description: there were no adverse events.
Groups:
- Clopidrogel + Aspirin: Single loading doses of Clopidogrel (600 mg) and ASA (325 mg), followed by daily dosing for 5-7 days (clopidogrel 75 mg + ASA 81 mg once daily).
Arm/Group | Ticagrelor + Aspirin | Clopidrogel + Aspirin
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes